CLINICAL TRIAL: NCT04230447
Title: Peking Union Medical College Hospital
Brief Title: Establishment of a Cohort of Patients With Sepsis-associated Encephalopathy (SAE)
Acronym: SAE
Status: Recruiting | Type: Observational
Sponsor: Yi Li, MD (Other)
Responsible Party: Sponsor-Investigator, Yi Li, MD, director billliyi@126.com, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: ZS-2165
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Sepsis-Associated Encephalopathy
Keywords: Sepsis-associated encephalopathy
MeSH Terms: conditions — Sepsis-Associated Encephalopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We are collecting the samples of the included participants, including whole blood, plasma, serum, cerebrospinal fluid, stool and rectal swabs.After the sample collection, the RNA-sequence, metabolites and cytokines were under detection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- sepsis associated encephalopathy (SAE): This study is an observational study without drug and other interventions The SAE was defined as the Glasgow Coma Scale (GCS) score of less than 15
  Interventions: Other: No intervention
- Non-SAE: This study is an observational study without drug and other interventions Non-SAE group GCS = 15
  Interventions: Other: No intervention
- Control: This study is an observational study without drug and other interventions The control group was the emergency department patients with acute disease strikes, including heart attack, infraction, and healthy control.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
In this study, the researcher involved the sepsis patients(defined by sepsis 3.0) in Peking Union Medical College Hospital. The SAE was defined as the Glasgow Coma Scale (GCS) score of less than 15 and the Non-SAE group GCS = 15. The control group was the non-infectious patients with acute disease strikes and the healthy control. After the sample collection, the RNA-sequence, metabolites and cytokines were under detection.

DETAILED DESCRIPTION:
We conducted a prospective observational cohort study of critically ill patients admitted to Emergency Department at a tertiary care hospital. This clinical study was approved by the Ethics Institutional Review Board of Peking Union Medical College Hospital. We identified the sepsis patients according to the Sepsis 3.0 criteria. The SAE was defined as the Glasgow Coma Scale (GCS) score of less than 15 and the Non-SAE group GCS = 15. The control group was the non-infectious patients with acute disease strikes and the healthy control.

We are collecting the samples of the included participants, including whole blood, plasma, serum, cerebrospinal fluid, stool and rectal swabs. The total RNA was extracted from the whole blood by PAXgene Blood RNA MDx kit (PreAnalytiX) for RNA sequence. We used the Ultra-high performance liquid chromatography-MS/MS (UHPLC-MS/MS) analysis for detected metabolites.

We used the Bio-Plex 200 system (Luminex Corporation, Austin, TX, USA) and Simoa HD-X AnalyzerTM (Quanterix) platform to detect cytokines.

ELIGIBILITY:
Inclusion criteria:

1. sepsis 3.0 diagnostic criteria;
2. Estimated length of hospital stay> 24h;
3. ages 18-89;
4. Acute brain dysfunction: delirium, coma, epilepsy, focal neurological deficit;
5. Patients who meet the non-infectious SIRS diagnostic criteria

Exclusion criteria:

1. Diagnosis of patients with brain injury before admission, including Alzheimer's disease, craniocerebral injury, etc .;
2. Primary brain injury (cerebral hemorrhage, cerebral infarction, etc.), secondary brain injury (liver brain, lung brain, uremia encephalopathy, pancreatic encephalopathy, metabolic encephalopathy, Wake encephalopathy, etc.);
3. pregnant and lactating women;
4. Those who have undergone bypass surgery in the past 3 months;
5. Hearing and vision impairment;
6. mental illness and melanoma;
7. Abnormal coagulation, active bleeding
8. Patients with infection at lumbar puncture site
9. Meningeal leukemia patients
10. Patients with other types of encephalopathy

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Meet the above three categories of patients consistent with inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2030-01-14 (Estimated)

PRIMARY OUTCOMES:
Finding the pathogenesis of sepsis encephalopathy | 2020-2030
  To find the pathogenesis of sepsis encephalopathy by genetic testing of blood and cerebrospinal fluid in patients with sepsis and sepsis and SIRS by molecular biomarkers and physiological parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qin M, Yu S, Lu X, Gong C, Song Z, Zhu H, Gao Y, Li Y. Reduced phosphatidylcholine and phosphatidylethanolamine levels correlate with inflammatory activation in sepsis-associated encephalopathy. Eur J Med Res. 2025 Aug 31;30(1):828. doi: 10.1186/s40001-025-03115-z. PMID 40887666